CLINICAL TRIAL: NCT00944554
Title: Relapse Prevention With Varenicline
Acronym: 0815
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NA_00019900
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-07

CONDITIONS: Recurrence; Smoking Cessation; Substance-Related Disorders
Keywords: Relapse; Smoking Cessation; Substance Abuse
MeSH Terms: conditions — Recurrence; Smoking Cessation; Substance-Related Disorders | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Group given placebo.
  Interventions: Drug: Placebo
- Varenicline (Experimental): Experimental group given varenicline dosing.
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline given twice a day or five weeks.
  Other Names: Varenicline (Chantix®)
  Arms: Varenicline
Drug: Placebo — Placebo given twice a day or five weeks.
  Arms: Placebo

SUMMARY:
This study aims to determine if varenicline (Chantix®), currently used as a smoking cessation aid, will decrease the likelihood of relapse to smoking following a programmed lapse in the laboratory. The hypothesis is that varenicline will reduce the reinforcing effects of smoking and will delay or prevent relapse compared to placebo.

DETAILED DESCRIPTION:
In this study, the investigators plan to use an experimental model of a lapse, in which volunteers smoke two cigarettes after a brief period of (12-24 hours). The goals of this study are to assess the impact of varenicline on the subjective and reinforcing effects of cigarettes, as well as the latency to resume smoking (relapse) following the lapse exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old
* Reports smoking at least 10 cigarettes per day AND provides a urine sample that tests positive for nicotine metabolites at intake
* Contemplating a smoking cessation attempt in the near future
* Willing to engage in a practice quit attempt during which they will be asked to smoke on one occasion
* Able to give informed consent

Exclusion Criteria:

* Currently meets Diagnostic and Statistical Manual (DSM-IV) criteria for depression, bi-polar disorder, or schizophrenia
* History of attempted suicide or expresses any current suicidal ideation
* Pregnant, breast feeding, or planning to become pregnant within the next 3 months
* Reports desire for immediate treatment of tobacco/nicotine dependence
* Severe impairment of renal function indicated by Glomerular Filtration Rate (GFR) less than 30 ml/min calculated using the Cockcroft and Gault prediction method (plasma creatinine adjusted by weight, gender, and age)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maxine L Stitzer, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Group given placebo twice a day for 5 weeks.
- Varenicline: Experimental group given varenicline twice a day or five weeks.
Period: Overall Study
Arm/Group | Placebo | Varenicline
Started | 50 | 54
Completed | 22 | 25
Not Completed | 28 | 29

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Group given placebo.
  Placebo: Varenicline and placebo given twice a day or five weeks.
- Varenicline: Experimental group given varenicline dosing.
  Varenicline: Varenicline and placebo given twice a day or five weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Varenicline | Total
Number analyzed (Participants) | 50 | 54 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (10) | 45 (12) | 44 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 32 | 52
  Male | 30 | 22 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 50 | 54 | 104
Region of Enrollment [Number; unit: participants]
  United States | 50 | 54 | 104

OUTCOME MEASURES:

1. Primary Outcome: Days to Relapse
Description: Number of days following the programmed lapse exposure until relapse to smoking occurred
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: days
Groups:
- Placebo: Group given placebo twice a day or five weeks.
Arm/Group | Placebo | Varenicline
Number analyzed (Participants) | 22 | 25
days | 9.1 (9.7) | 16.4 (10.3)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Placebo | Varenicline
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/54
Other Adverse Events (participants affected / at risk) | 0/50 | 0/54

LIMITATIONS AND CAVEATS:
Experimental model of relapse used in non-treatment seeking smokers. Results may not generalize to all smokers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No